CLINICAL TRIAL: NCT01255917
Title: Nerve Growth Factor in Chronic Pancreatitis
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: HM11033
Record Dates: First submitted 2010-12-06; First posted 2010-12-08 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Pancreatitis
Keywords: Tio identify role of NGF in pain in CP; Identify biomarkers related to progression of CP
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pancreatic fluid obtained by duodenal aspiration
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic pancreatitis

SUMMARY:
This study is to understand the role of nerve growth factor(NGF) and other cytokines in the pancreatic fluid of patients with chronic pancreatitis.

Hypothesis:

1. Pain does not correlate with changes in the PD morphology suggesting that pain in CP is not only a mechanical problem
2. Pain in CP correlates better with the levels of NGF in the pancreatic juice. NGF is variably expressed in different morphological stages of CP and regulates the sensitivity of the peptidergic nociceptors and is upregulated in pancreatic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established CP and none of the exclusion criteria mention below.

Exclusion Criteria:

* Failure to obtain consent.
* Any comorbid condition with expected survival < 1 year.
* Patients with pacemaker, implanted metallic prosthesis or other contraindications to do MRCP.
* Patients < 18 years of age at time of consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Test group: Subjects with CP in each morphological stage and matched for age, race, gender, narcotic dependence and etiology of CP will be enrolled Controls: Subjects undergoing upper gastrointestinal endoscopy (UGIE) for non-pancreatic causes.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2008-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The levels of NGF in subjects with different morphological stages of chronic pancreatitis (CP) will be compared to the controls and in each morphological stage of CP will be correlated with pain scores. | 5 years

SECONDARY OUTCOMES:
Correlate the expression of NGF and other inflammatory cytokines in the pancreatic juice in each morphological stage of CP. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bimaljit S Sandhu, M.D, Principal Investigator — Associate Professor, VCU Medical Center
Locations (1):
- Virginia Commonwealth University Medical Center, Richmond, Virginia, United States